CLINICAL TRIAL: NCT00231946
Title: A Double-Blind Placebo-Controlled Study of VP4896 For the Treatment of Mild-to-Moderate Alzheimer's Disease
Brief Title: ALADDIN Study - Phase III: Antigonadotropin-Leuprolide in Alzheimer's Disease Drug INvestigation (VP-AD-301)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Voyager Pharmaceutical Corporation (Industry)
Organization: National Institute on Aging (NIA) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IA0084
Record Dates: First submitted 2005-09-30; First posted 2005-10-04 (Estimated); Last update posted 2007-09-20 (Estimated); Status verified 2007-09

CONDITIONS: Alzheimer's Disease
Keywords: gonadotropins; hormone therapy; HRT; Antigonadotropin; Leuprolide
MeSH Terms: conditions — Alzheimer Disease

INTERVENTIONS:
Drug: VP4896

SUMMARY:
The study is designed to investigate the activity of the hormone drug leuprolide acetate in stabilizing cognitive function in mild-to-moderate AD patients.

DETAILED DESCRIPTION:
VP4896 is a gonadotropin releasing hormone (GnRH) agonist that binds to and inactivates GnRH receptors on the pituitary gland. This decreases the amount of luteinizing hormone released by the pituitary. The hypothesis upon which this trial is designed is that luteinizing hormone is the cause of Alzheimer's disease. VP4896 decreases the amount of luteinizing hormone in the body and, therefore, may decrease or halt the progression of Alzheimer's disease.

This is a double-blind, placebo-controlled, study designed to assess the safety and efficacy of VP4896 (a novel formulation of leuprolide acetate) in the treatment of subjects with mild-to-moderate AD. The study duration is 56 weeks. Approximately 555 participants will be recruited from approximately 80 sites in the United States, Canada, and South America.

The study drug will be administered every eight weeks over a 48 week period. Male subjects randomized to active treatment will also receive testosterone replacement gel.

The change from baseline in ADAS-Cog (cognitive test) score at Week 50 and ADCS-CGIC (global cognitive and behavioral measure) at Week 50 will be the primary efficacy endpoints. Safety will be assessed at all visits and by phone at Week 1.

ELIGIBILITY:
Inclusion Criteria:

* 60 years of age or older
* Diagnosis of probable mild-to-moderate Alzheimer's Disease
* On a stable dose of an acetylcholinesterase inhibitor (including, but not limited to: donepezil, galantamine, rivastigmine, and tacrine) for at least 120 days prior to baseline and will likely remain on the drug throughout the trial; all participants must be on acetylcholinesterase inhibitors
* No other significant or interfering medical conditions

Exclusion Criteria:

* Significant neurological disease affecting the brain or psychiatric disease other than AD, such as current untreated major depression, schizophrenia, epilepsy, Parkinson's disease, Creutzfeldt-Jakob's disease, or clinical episode of stroke
* Laboratory or clinical signs of untreated, clinically significant abnormal thyroid function, in the Investigator's opinion
* Received other investigational drugs within 30 days or 5 half-lives prior to baseline, whichever is longer
* Taking other medications, with the exception of estrogen, known to affect serum gonadotropin (Gn) concentrations, including but not limited to goserelin, danazol, or leuprolide
* Other exclusion criteria exist--eligibility can be assessed by the trial site

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 555
Dates: Start 2005-09

PRIMARY OUTCOMES:
Cognitive assessment and Caregiver's impression of change at baseline and at weeks 8, 24, 34, and 50.

SECONDARY OUTCOMES:
Ability to perform Activities of Daily Living (ADL) at baseline and weeks 8, 24, 34, and 50. Impression of disease severity assessment at week 50.

CONTACTS AND LOCATIONS:
Overall Officials: Connie Powers, Principal Investigator — Sr. Clinical Scientist, Voyager Pharmaceutical
Locations (59):
- United States (55):
  - Pivotal Research Centers, Peoria, Arizona
  - NeuroSpecialists, PLLC, Tucson, Arizona
  - Margolin Brain Institute, Fresno, California
  - Bay Area Research Institute, Lafayette, California
  - Anderson Clinical Research, Loma Linda, California
  - Pharmacology Research Institute, Los Alamitos, California
  - David Trader, Los Angeles, California
  - Synergy Clinical Research, National City, California
  - Pharmacology Research Institute, Newport Beach, California
  - Pharmacology Research Institute, Northridge, California
  - North County Neurology Assoc., Oceanside, California
  - Pharmacology Research Institute, Riverside, California
  - Pacific Research Network, San Diego, California
  - San Francisco Clinical Research Center, San Francisco, California
  - Neurological Research Institute, Santa Monica, California
  - Torrance Clinical Research, Torrance, California
  - Radiant Research, Denver, Colorado
  - Colorado Neurology & Headache Center, Denver, Colorado
  - Comprehensive Neuroscience, Inc., Darien, Connecticut
  - Geriatric and Adult Psychiatry, Hamden, Connecticut
  - Meridien Research, Brookville, Florida
  - Brain Matters Research, Delray Beach, Florida
  - Berma Research Group, Hialeah, Florida
  - Neurology Clinical Research, LLC, Plantation, Florida
  - Roskamp Institute, Sarasota, Florida
  - Meridien Research, St. Petersburg, Florida
  - Meridien Research, Tampa, Florida
  - Palm Beach Neurological Group, West Palm Beach, Florida
  - Quantum Laboratories, West Palm Beach, Florida
  - Kuakani Medical Center, Honolulu, Hawaii
  - Booker, J. Gary, MD, APMC, Shreveport, Louisiana
  - ICPS Group, Boston, Massachusetts
  - Pivotal Research Centers, Royal Oak, Michigan
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Hunterdon Medical Center, Flemington, New Jersey
  - Albuquerque Neuroscience Inc., Albuquerque, New Mexico
  - Upstate Clinical Research, LLC, Albany, New York
  - Medark Clinical Trials, Morgantown, North Carolina
  - Raleigh Neurology Associates, P.A., Raleigh, North Carolina
  - Piedmont Medical Research Associates, Winston-Salem, North Carolina
  - Ohio State University Medical Center, Columbus, Ohio
  - Neurology Center of Ohio, Toledo, Ohio
  - IPS Research Company, Oklahoma City, Oklahoma
  - Pharmaceutical Research-Oregon, Inc., Eugene, Oregon
  - Clinical Trial Center, LLC., Jenkintown, Pennsylvania
  - Pearl Clinical Research, Inc., Norristown, Pennsylvania
  - Memory Research Institute, East Providence, Rhode Island
  - Butler Hospital, Providence, Rhode Island
  - Norman Gordon, MD, Providence, Rhode Island
  - Radiant Research - Greer, Greer, South Carolina
  - University of Texas Health Science Center at Houston, Houston, Texas
  - Bexar Diagnostic Medicine Associates, San Antonio, Texas
  - Grayline Clinical Drug Trials, Wichita Falls, Texas
  - Southwestern Vermont Medical Center, Bennington, Vermont
  - Innovative Clinical Research Center, Alexandria, Virginia
- Canada (4):
  - The Medical Arts Health Research Group, Penticton, British Columbia
  - Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - Toronto Memory Program (Neurology Research Inc.), Toronto, Ontario
  - Novabyss Inc., Sherbrooke, Quebec

REFERENCES:
- [Background] Gregory CW, Bowen RL. Novel therapeutic strategies for Alzheimer's disease based on the forgotten reproductive hormones. Cell Mol Life Sci. 2005 Feb;62(3):313-9. doi: 10.1007/s00018-004-4386-y. PMID 15723167
- [Background] Bowen RL, Atwood CS. Living and dying for sex. A theory of aging based on the modulation of cell cycle signaling by reproductive hormones. Gerontology. 2004 Sep-Oct;50(5):265-90. doi: 10.1159/000079125. PMID 15331856
- [Background] Bowen RL, Verdile G, Liu T, Parlow AF, Perry G, Smith MA, Martins RN, Atwood CS. Luteinizing hormone, a reproductive regulator that modulates the processing of amyloid-beta precursor protein and amyloid-beta deposition. J Biol Chem. 2004 May 7;279(19):20539-45. doi: 10.1074/jbc.M311993200. Epub 2004 Feb 9. PMID 14871891
- [Background] Webber KM, Bowen R, Casadesus G, Perry G, Atwood CS, Smith MA. Gonadotropins and Alzheimer's disease: the link between estrogen replacement therapy and neuroprotection. Acta Neurobiol Exp (Wars). 2004;64(1):113-8. doi: 10.55782/ane-2004-1497. PMID 15190686
- [Background] Zhu X, McShea A, Harris PL, Raina AK, Castellani RJ, Funk JO, Shah S, Atwood C, Bowen R, Bowser R, Morelli L, Perry G, Smith MA. Elevated expression of a regulator of the G2/M phase of the cell cycle, neuronal CIP-1-associated regulator of cyclin B, in Alzheimer's disease. J Neurosci Res. 2004 Mar 1;75(5):698-703. doi: 10.1002/jnr.20028. PMID 14991845
- See also: Alzheimer's Disease Education and Referral Center — http://www.alzheimers.org
- See also: Alzheimer's Association — http://www.alz.org